CLINICAL TRIAL: NCT06315478
Title: Safety and Efficacy of Triple and Quadruple Regimens as First Line Therapy for Management of Helicobacter Pylori Infection in Egyptians
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Donia Mohamed Eid, bachelor graduate at pharmacy university, Helwan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Hybrid regimen for H.pylori
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: H.Pylori Infection
MeSH Terms: interventions — Omeprazole; Tablets; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple regimen(Group A) (Active Comparator)
  Interventions: Drug: Omeprazole 20 MG Oral Tablet
- Quadruple regimen (Group B) (Active Comparator)
  Interventions: Drug: Amoxicillin 500Mg Tab
- Hybrid regimen (Group C) (Active Comparator)
  Interventions: Drug: Clarithromycin 500Mg Tab

INTERVENTIONS:
Drug: Omeprazole 20 MG Oral Tablet — standard triple therapy for 14 days Bid for each drug
  Other Names: amoxicillin 500 mg; clarithromycin 500mg
  Arms: Triple regimen(Group A)
Drug: Amoxicillin 500Mg Tab — Quadruple regimen for 14 days Bid for each drug
  Other Names: Omeprazole 20 MG Oral Tablet; clarithromycin 500mg; metronidazole 500mg
  Arms: Quadruple regimen (Group B)
Drug: Clarithromycin 500Mg Tab — Hybrid regimen, PPI and Amoxicillin for first 7 days then adding clarithromycin and metronidazole for the second 7 days
  Other Names: amoxicillin 500 mg Tablet; Omeprazole 20 MG Oral Tablet; metronidazole 500mg Tablet
  Arms: Hybrid regimen (Group C)

SUMMARY:
Our study aimed to investigate the efficacy and safety of hybrid regimen as a first line therapy for H. pylori eradication compared to triple and quadruple regimens in attempt to overcome antibiotic resistance

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) is a globally prevalent pathogen which infects about over 50% of population. However, not all cases have clinical symptoms, H. pylori are described as gram negative bacteria which causes ulcers in the lining of stomach or the upper part of small intestine. For some patients, a progressive infection can cause gastric cancer which is the second widespread cancer worldwide (1).

While this pathogen in Egypt is a public health issue, the propagation of H. pylori infection is approximately 80% (2), study results concluded that H. pylori infection in upper Egypt was higher than in urban areas (3).

Transmission modes of H. pylori are very controversial, the reservoir of H. pylori is the human stomach. The main method of acquisition in both developing and developed countries by fecal oral route, whereas the other route of transmission in developed countries is the gastro-oral route mainly water borne prevalence, overcrowding of the family of large number members, institutionalized children are predisposing for acquiring the infection. (4:6), and occupational risk factor for health members, in particular those working in gastrointestinal units (7). Over spread of the infection in upper Egypt could be due to the hygiene level, socioeconomic conditions, life style, and absence of sources of pure water supply in rural areas (3).

H. pylori has been classified as one of the 12 bacterial species need high priority future strategies for new antibiotic development by the World Health Organization (WHO), management of H. pylori is widely debatable due to high antibiotics resistance prevalence after exclusion of inadequate gastric suppression by proton pump inhibitor and poor adherence to the therapy. Furthermore, the efficacy of many regimens has declined due to increased antibiotic resistance making H. pylori eradication challenging, H. pylori treatment has been complicated and has required 10 and 14 days of multiple daily doses of three or four different medicines. (8:13).

There is no worldwide accepted regimen for the eradication of H. pylori infection. Standard triple therapy (STT) with proton pump inhibitors (PPI) in standard dose, clarithromycin (500 mg), and amoxicillin (1 g) twice daily for 14 days is the standard triple first line regimen in the published international guidelines of the European Helicobacter and Microbiota Study Group in areas of low clarithromycin resistance (14).

A randomized controlled trial in Japan showed that clarithromycin resistance is a growing problem found metronidazole to be superior to clarithromycin as a 7-day first-line triple regimen (15).

In regions with low dual clarithromycin and metronidazole resistance (<15%), either a bismuth quadruple therapy (BQT) (PPI, bismuth salt, tetracycline, and metronidazole) or non-bismuth concomitant quadruple therapy (PPI, amoxicillin, clarithromycin, and metronidazole) is recommended (14,16), In areas of high dual clarithromycin and metronidazole resistance (>15%), bismuth quadruple therapy is the recommended regimen. However, bismuth isn't available in all regions and not preferred due to complexity and the high pill burden (14 pills per day). Therefore, levofloxacin, rifabutin or high dose dual (amoxicillin and PPI) therapies have been suggested (14,17).

A levofloxacin triple therapy is recommended as second-line treatment in case of first line therapy failure; However, clarithromycin-based triple therapy or bismuth quadruple therapy are alternative second-line options if not used as first line regimen and clarithromycin resistance is known to be low.

Third-line and subsequent treatment strategies should be guided by antimicrobial susceptibility testing, treatment durations of 14 days and the use of newer generation PPIs are recommended in all H. pylori regimens, unless local evidence suggests that 10 days therapy is efficient (14,18,19). In Egypt, the first and second line H. pylori regimens as the international guidelines are used to eradicate H.pylori. However, these recommendations should be reviewed, due to increased resistance rate and progressive decline in eradication therapy efficacy. (20).

Expert groups in USA, Canada, and Europe have issued treatment guidelines for the management of H. pylori infection to overcome the global challenge of antibiotic resistance (13).

Treatment of H. pylori is still widely empiric due to antibiotic resistance, which could be prevented through culture guided therapy that associated with higher eradication rates (21,22).

Some experts such as the Maastricht guidelines recommend clarithromycin susceptibility testing before prescribing clarithromycin triple regimen or after second line regimen failure, its preferable to have this test in an earlier phase than waiting for two treatment failures mostly due to increased levofloxacin resistance, a component of many second line therapies (14,23,24).

Antibiotic susceptibility testing can be done by culture or molecular methods, both of which require gastric biopsies. However. This test is less cost-effective to be adopted widespread (23). The scarcity of such data in USA was an obstacle to make strong evidence-based treatment recommendations in the 2017 ACG guideline on H. pylori treatment (19).

In USA, only two publications in the previous 20 years including fewer than 500 strains of H. pylori have revealed resistance features (13,25,26) A recent study compared the efficacy of first-line H.pylori eradication therapies including STT, BQT, sequential therapy (ST) consisting of a PPI and amoxicillin for 5-7 days followed by a PPI, clarithromycin, and a metronidazole for 5-7 days, and HT. Results revealed that hybrid regimen had the best H.pylori eradication rates (27).

Another study compared the efficacy of different regimens for eradication of H. pylori had shown that A 14-day hybrid therapy has attracted global attention as this regimen proved to be safe, well tolerated and effective in high antibiotic resistance settings (28,29).

A current hybrid therapy (HT) (PPI and amoxicillin for 14 days followed by clarithromycin and a nitroimidazole for 7 days) is a promising first-line strategy for H. pylori eradication due to the rising prevalence of antibiotic resistance globally (30).

To the best of our knowledge there is lacking information about hybrid regimen efficacy in eradication of H.pylori infection in Egyptian patients, our study aimed to investigate the efficacy and safety of hybrid regimen as a first line therapy for H. pylori eradication compared to triple and quadruple regimens in attempt to overcome antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria:

* 1. Naïve patients 2. adult >18 years 3. Patients with positive SAT 4. Patients didn't take any antibiotics for the previous 4 weeks or PPI for the previous 2 weeks 5. Patients diagnosed with duodenal ulcers who have H. pylori infection and treated with triple or quadruple regimens for H. pylori

Exclusion Criteria:

* 1-Patients had any concern with triple or quadruple regimens such as hypersensitivity to any of the drug 2-Pregnancy or lactation 3-Refusal to sign the informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
stool antigen retest | 6 weeks
  efficacy of the regimen by eradication of H. pylori

CONTACTS AND LOCATIONS:
Locations (1):
- Badr hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No